CLINICAL TRIAL: NCT03453411
Title: Multicentre, Prospective, Uncontrolled Study to Describe the Present, Felt and Sought Effects of EMONO in Children During Dental Care
Brief Title: Effects of EMONO in Children During Dental Care
Acronym: MEOPAeDent
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Agence Nationale de sécurité du Médicament (Other)
Responsible Party: Sponsor
Other Study IDs: RC17_0421
Record Dates: First submitted 2018-02-26; First posted 2018-03-05 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2018-02

CONDITIONS: Dental Care
Keywords: Equimolar Mixture of Oxygen and Nitrous Oxide (EMONO); Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non interventional study
  Interventions: Other: Non interventional study

INTERVENTIONS:
Other: Non interventional study — Non interventional study

SUMMARY:
The main objective of this project is to evaluate the effects sought and the effects felt by children when EMONO is used in pediatric dental care. The Investigators will try to characterize the children who have submitted a request to extend contact with EMONO. The maintenance of a framework for the safe use of this drug whose place in dental care is fundamental and the benefit ratio is very favorable is essential.

DETAILED DESCRIPTION:
Some narcotic drugs and psychotropic drugs associated with a risk of misuse or identified dependence and are, moreover, the object of a reinforced surveillance. This is the case of EMONO (Equimolar Oxygen and Nitrogen Protoxide Mix), which is part of the ANSM (French National Agency for Medicines and Health Products Safety) list of drugs with enhanced surveillance. EMONO is a gas composed equally of oxygen and nitrous oxide (also called laughing gas). He has had a marketing authorization in France since 2001. Until 2009, it was reserved for hospital use. Since 2009, a modification of its MA has enabled the release of the hospital reserve, EMONO can now be used in city medicine and dental surgery. The ANSM has made its provision outside health facilities conditional on the implementation of a common national RMP, accompanied by a national monitoring of pharmacovigilance and addictovigilance. The latter is under the responsibility of CEIP-A of Nantes.

The use of EMONO in pediatric dental care is a particular mode of use in a pediatric population in which the administration of EMONO is often the first administration of a psychoactive substance known for its positive effects (euphoria). Health professionals daily observe children, who after care under EMONO, have a strong appetite for EMONO and claim for any intervention. It would be necessary to understand why, and to estimate the number of children involved. Do children feel positive effects during these actions, which could lead to a wish to prolong the contact with the gas, in search of an effect other than therapeutic? The main objective of this project is to evaluate the effects sought and the effects felt by children when EMONO is used in pediatric dental care. The investigators will try to characterize the children who have submitted a request to extend contact with EMONO. The maintenance of a framework for the safe use of this drug whose place in dental care is fundamental and the benefit ratio is very favorable is essential.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 15, requiring care under MEOPA

Exclusion Criteria:

* Do not fit into the inclusion criteria

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: For this study we have therefore chosen to include all patients under 15 years of age seen for care under EMONO in the different participating DSCs. The use of EMONO in dental care is indicated for minor patients who are not cooperating in the dental care (doing not allow the realisation in the chair of care according to the acquired data of science) or who have a handicap limiting their cooperation. It applies during diagnostic or therapeutic consultations. The investigators will not include patients under 3 years of age as EMONO is much less effective below this age. All dental surgeons of the participating DSCs will be responsible for selecting patients who meet the inclusion criteria, offering selected patients and their parents to participate and include them in the study.
Sampling Method: Probability Sample
Enrollment: 679 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2020-06-24 (Actual)

PRIMARY OUTCOMES:
Description of the effects felt and sought after by EMONO during the first care session. | Day 0
  Exhaustive interview of patients about the presence or absence of each expected effect of EMONO and each adverse event at the first session of care; with also questioning the perception of this effect (positive or not).

SECONDARY OUTCOMES:
Assess the child's appreciation of the EMONO | Day 0
  VAS score of contact with EMONO
Characterization of children who experience both analgesia and anxietyolysis | Day 0
  Choice of the child (inhalation of EMONO) with the minting tool test (drug-liking)
Evaluate children's palatability for EMONO and characterize children with high palatability. | Day 0
  Composite criterion
Evaluate the course of taking EMONO between the first and the last session of care | Month 1
  Evolution of the effective dose between the first and last treatment session
Assess the impact of the difference in practice between the French University Hospitals on anxiety | Day 0
  Composite criterion

CONTACTS AND LOCATIONS:
Overall Officials: Tony Prud'homme, Dr, Principal Investigator — Nantes University Hospital
Locations (1):
- Chu de Nantes, Nantes, France

REFERENCES:
- [Derived] Prud'homme T, Rousselet M, Istvan M, Cheraud-Carpentier M, Dajean-Trutaud S, Lopez S, Muller-Bolla M, Marty M; French Pediatric Dentistry Network (FPDN); Feuillet F, Victorri-Vigneau C. Equimolar oxygen-nitrous oxide (EMONO) in dental pediatric care: which patients achieve therapeutic effects? A French national exploratory prospective observational multicenter study. Eur Arch Paediatr Dent. 2025 Feb;26(1):149-158. doi: 10.1007/s40368-024-00950-2. Epub 2024 Nov 15. PMID 39548019
- [Derived] Prud'homme T, Dajean-Trutaud S, Rousselet M, Feuillet F, Carpentier-Cheraud M, Bonnot O, Hyon I, Grall-Bronnec M, Lopez-Cazaux S, Victorri-Vigneau C. The MEOPAeDent trial protocol-an observational study of the Equimolar Mixture of Oxygen and Nitrous Oxide (EMONO) effects in paediatric dentistry. BMC Oral Health. 2019 Mar 7;19(1):42. doi: 10.1186/s12903-019-0732-6. PMID 30845960